CLINICAL TRIAL: NCT05856253
Title: Implementation and Early Results on an Enhanced Recovery Program in Esophageal Surgery
Brief Title: Enhanced Recovery in Esophageal Surgery
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Deswysen Yannick, Chef de Clinique Associé, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2023/23Jan/038
Record Dates: First submitted 2023-04-07; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: ERAS Protocol, Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group
  Interventions: Procedure: Enhanced recovery program
- Control group

INTERVENTIONS:
Procedure: Enhanced recovery program — Recvoery programs includes specific measures validated in multidisciplinary consultation, spread over the pre- intra- and postoperative period.
  Groups: ERAS group

SUMMARY:
Esophageal surgery remains the main treatment for esophageal cancer. Despite constant improvements, morbidity of esophagectomy remains high. For several years, enhanced rehabilitation programs have been used to reduce the impact of surgery on the patients to support a faster recovery. This study analyses the first results of newly implemented enhanced program after esophagectomy within the framework of an academic center.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive esophagectomy

Exclusion Criteria:

* Contraindication for surgery according to the WHO physical status of IV, emergency surgery, mental illness and patient's refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients operated on esophagectomy for malignant and non malignant esophageal pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who reach the the 23 measurements of the enhanced recovery program | an average of 15 days (During the surgical period (hospital stay)
  compliance is defined by the achievement of the various items of the rehabilitation program (23 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No